CLINICAL TRIAL: NCT03607721
Title: Accuracy of Markerless 3D Motion Capture Evaluation to Differentiate Between On/Off Status in Parkinson's Disease After Deep Brain Stimulation
Brief Title: Accuracy of Markerless Motion Capture Evaluation in Parkinson's Disease After DBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Zambrano Hellion (Other)
Responsible Party: Principal Investigator, Hector Ramon Martinez, Director of Instituto de Neurologia y Neurocirugia Hospital Zambrano Hellion, Hospital Zambrano Hellion
Organization: INNCMZH (Unknown)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DARI-DBS
Record Dates: First submitted 2018-07-04; First posted 2018-07-31 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Parkinson Disease
Keywords: deep brain stimulation; kinematics; markerless; body motion evaluation; gait analysis
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Participants were divided in two groups: Parkinson's Disease patients that underwent deep brain stimulation and a control group with healthy subjects matched by age and gender.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DBS Patients Group (Experimental): Body Motion Evaluation DARI
  Interventions: Device: Body Motion Evaluation DARI
- Control Group (Active Comparator): Body Motion Evaluation DARI
  Interventions: Device: Body Motion Evaluation DARI

INTERVENTIONS:
Device: Body Motion Evaluation DARI — Dynamic Athletic Research Institute (DARI) Software to evaluate motion tridimensionally with a camera system and without the use of body sensors.

SUMMARY:
Body motion evaluation (BME) by markerless systems is increasingly being considered as an alternative to traditional marker-based technology because they are faster, simpler, and less expensive. They are increasingly used in clinical settings in patients with movement disorders, however, the wide variety of systems available make results conflicting.

The objective of this study was to determine if a markerless 3D motion capture system is a useful instrument to objectively differentiate between Parkinons's Disease (PD) patients with Deep Brain Stimulation (DBS) in On and Off state and controls; and its correlation with the evaluation by means of Unified Parkinson's Disease Rating Scale (UPDRS).

Six PD patients who underwent DBS bilaterally in the subthalamic nucleus were evaluated using BME and UPDRS-III with DBS turned On and Off. BME of 16 different movements in six controls paired by age and sex was compared with PD patients with DBS in On and Off states.

Kinematic data obtained with this markerless system could contribute to the discrimination between PD patients and healthy controls. This emerging technology may help to clinically evaluate PD patients more objectively.

DETAILED DESCRIPTION:
Methodology. Patients. Six patients with PD, diagnosed in accordance with the United Kingdom Parkinson's Disease Society Brain Bank Clinical Diagnostic Criteria by a certified neurologist and movement disorder specialist, were included. This is a pilot study, and sample size was chosen by convenience, accessibility and proximity to the researchers. The study was approved by the investigator's institutional research board, and the patients and controls provided written consent. In the months preceding the test, the PD patients were clinically evaluated by the same physician according to the Unified Parkinson Disease Rating Scale section III or motor section (UPDRS-III).

Instrument. Actually, there are many markerless motion capture systems in the market, with a broad range of prices, as well as a broad range of reliability. However, DARI system has been proven to be one of the best for numerous reasons. This system requires a quick calibration at the beginning of each day that the technician can complete in less than 10 minutes. It does not have to be repeated until the following day, no matter how many patients are evaluated. The system depends on a computer-based software that acquires the patient's skeleton or avatar using eighteen high-speed cameras (120 Hz) placed around the room to collect whole body data and delivers kinematic analysis almost instantly using sophisticated biomechanical algorithms.

Also, traditional motion labs use cumbersome floor-mounted pressure plates to measure the forces generated by the body. These require frequent calibration and restrict the subject's movement to a limited area. DARI's kinetic capture system does not require force plates and can measure joint torques, ground reaction forces, and other measurements without restricting the subject's natural movement.

Markerless 3D motion capture evaluation of kinematics in the PD patients and controls was performed on a rectangle room that measures 6 x 6 meters and 3 meters in height. The room has a green screen on the floor, and eighteen cameras are strategically placed on the walls, twelve are placed 2.6 meters high and 6 are on a lower level at 30 centimeters from the ground. The room has ample space, which allows for broader movements to be analyzed.

Evaluations. PD patients were asked to arrive in the morning wearing dark close-fitting clothing, to skip their last PD medication, and with DBS in Off state for least 180 minutes. On PD patients, UPDRS-III evaluation was done first. Then, to begin the markerless body motion evaluation (BME), patients and controls' weight and height were entered into the system to help establish the locations of joint centers. Once inside the green room, subjects first stood with feet apart and arms outstretched to the side, while the system created a 3D silhouette of each participant's form and a biometric skeleton was acquired; this took no more than three seconds. For the BME, all subjects performed 16 different movements. This set of movements was especially designed to evaluate PD patients and contains items that are related to three major motor symptoms in this disease: rigidity, bradykinesia and postural instability; tremor is not possible to assess. Once the BME was done, PD patients were asked to turn their DBS to On state and wait 30 minutes before repeating both UPDRS-III and BME. Controls only performed the BME, which took no more than 20 minutes. PD patients were evaluated twice (DBS state On and Off) with a 1-hour wait in between; their evaluation altogether took approximately 1.5 hours. The data files were uploaded to DARI Motion Platform where the biomechanical analysis produced full-body kinematic results and, finally, these data were exported to Excel for statistical analysis.

Analysis. A paired t-test was used to compare mean changes in UPDRS-III between the On and Off state. Mean differences between groups were evaluated with ANOVA or Kruskal-Wallis tests depending of the distribution of the data of each independent variable. Post hoc analyses were made for pairwise comparison in statistically significant results. Bivariate correlations among evaluation modalities were examined. These correlations were examined in the On and Off state between UPDRS-III and BME items. To compare them as accurately as possible, the items on UPDRS-III and BME that were similar were correlated (e.g. rigidity in upper limbs from UPDRS-III was correlated with shoulder flexion, extension, rotation from BME). One of the correlations was hip displacement taken from BME, which analyzes balance by measuring the movement of hips when patients stand during 10 seconds with arms outstretched to the sides and eyes closed; this was correlated with posture stability item from UPDRS-III, which is a quick pull, reactionary intervention test where patient's response is measured. Because not all UPDRS-III items were measurable by DARI, seven out of 18 were correlated; however, all BME items were correlated with UPDRS-III global score. IBM SPSS Statistics 21.0 software was used for data analysis. A p-value of ≤0.05 was considered to indicate statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Diagnosis of Parkinson's Disease by United Kingdom Parkinson's Disease Society Brain Bank Clinical Diagnostic Criteria
* Submitted to subthalamic DBS implantation a minimum of 3 months prior to the evaluation.

Exclusion Criteria:

* Patients with physical disability (i.e. wheelchair, cane, assistance to daily living activities)
* History of stroke and physical disability
* Another neurological disorder other than PD
* Recent head and limb trauma that limits movement
* Treatment with antipsychotics or recent botulinum toxin treatment.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Shoulder Flexion (right and left), Shoulder Extension (right and left), Internal Shoulder Rotation (right and left), External Shoulder Rotation (right and left), Maximum shoulder abduction (right and left) | 1 day: Test is done twice. First with DBS in Off state and then repeated 1 hour after DBS has been turned to On state.
  Measured by DARI Body Motion Analysis. Range of movement, measured in degrees.
Bilateral squat depth, Lunge Distance (right and left), Step Length (right and left), Step Width (right and left) | 1 day: Test is done twice. First with DBS in Off state and then repeated 1 hour after DBS has been turned to On state.
  Measured by DARI Body Motion Analysis. Range of movement, measured in centimeters.
Trunk Rotation, Trunk Flexion, Trunk Extension | 1 day: Test is done twice. First with DBS in Off state and then repeated 1 hour after DBS has been turned to On state.
  Measured by DARI Body Motion Analysis. Range of movement, measured in degrees.
Anterior-posterior hip displacement, Medial-lateral hip displacement | 1 day: Test is done twice. First with DBS in Off state and then repeated 1 hour after DBS has been turned to On state.
  Measured by DARI Body Motion Analysis. Patients are asked to outstretch their arms to the sides, extend their neck and close their eyes during 10 seconds. The hip displacement that happens during this time is recorded and measured in centimeters.
Cadence | 1 day: Test is done twice. First with DBS in Off state and then repeated 1 hour after DBS has been turned to On state.
  Measured by DARI Body Motion Analysis. Measured in steps/minute.
Speed or velocity | 1 day: Test is done twice. First with DBS in Off state and then repeated 1 hour after DBS has been turned to On state.
  Measured by DARI Body Motion Analysis. Measured in meters/second.
Stride length | 1 day: Test is done twice. First with DBS in Off state and then repeated 1 hour after DBS has been turned to On state.
  Measured by DARI Body Motion Analysis. It is the distance between any two successive points of heel contact of the same foot. Measured in centimeters.

SECONDARY OUTCOMES:
Speech | 1 day: Test is done once with DBS in Off state.
  Unified Parkinson's Disease Rating Scale Section III (motor examination). Score ranges from 0-4 where 0 is normal and 4 is unintelligible.
Facial Expression | 1 day: Test is done once with DBS in Off state.
  Unified Parkinson's Disease Rating Scale Section III (motor examination). Score ranges from 0-4 where 0 is normal and 4 is severe or complete loss of facial expression.
Tremor at Rest | 1 day: Test is done once with DBS in Off state.
  Unified Parkinson's Disease Rating Scale Section III (motor examination). Head, upper and lower extremities. Score ranges from 0-4 where 0 is absent and 4 is marked in amplitude and present most of the time.
Action or Postural Tremor of Hands | 1 day: Test is done once with DBS in Off state.
  Unified Parkinson's Disease Rating Scale Section III (motor examination). Score ranges from 0-4 where 0 is absent and 4 is marked in amplitude and interferes with feeding.
Rigidity | 1 day: Test is done once with DBS in Off state.
  Unified Parkinson's Disease Rating Scale Section III (motor examination). Judged on passive movement of major joints with patient relaxed in a sitting position. Score ranges from 0-4 where 0 is absent and 4 is severe, range of motion achieved with difficulty.
Finger Taps | 1 day: Test is done once with DBS in Off state.
  Unified Parkinson's Disease Rating Scale Section III (motor examination). Tapping of thumb and index finger in rapid succession. Score ranges from 0-4 where 0 is normal and 4 is can barely perform the task.
Hand Movements | 1 day: Test is done once with DBS in Off state.
  Unified Parkinson's Disease Rating Scale Section III (motor examination). Opening and closing hands in rapid succession. Score ranges from 0-4 where 0 is normal and 4 is can barely perform the task.
Rapid Alternating Movements of Hands | 1 day: Test is done once with DBS in Off state.
  Unified Parkinson's Disease Rating Scale Section III (motor examination). Pronation-supination in rapid succession. Score ranges from 0-4 where 0 is normal and 4 is can barely perform the task.
Leg Agility | 1 day: Test is done once with DBS in Off state.
  Unified Parkinson's Disease Rating Scale Section III (motor examination). Tapping heel on the ground in rapid succession picking up entire leg. Score ranges from 0-4 where 0 is normal and 4 is can barely perform the task.
Arising from Chair | 1 day: Test is done once with DBS in Off state.
  Unified Parkinson's Disease Rating Scale Section III (motor examination). Patient attempts to rise from straight-backed chair with arms folded across chest. Score ranges from 0-4 where 0 is normal and 4 is unable to arise without help.
Posture | 1 day: Test is done once with DBS in Off state.
  Unified Parkinson's Disease Rating Scale Section III (motor examination). Score ranges from 0-4 where 0 is normal, erect and 4 is marked flexion with extreme abnormality of posture.
Gait | 1 day: Test is done once with DBS in Off state.
  Unified Parkinson's Disease Rating Scale Section III (motor examination). Score ranges from 0-4 where 0 is normal and 4 is cannot walk at all, even with assistance.
Postural Stability | 1 day: Test is done once with DBS in Off state.
  Unified Parkinson's Disease Rating Scale Section III (motor examination). Response to sudden, strong posterior displacement produced by pull on shoulders while patient erect with eyes open and feet slightly apart. Score ranges from 0-4 where 0 is normal and 4 is unable to stand without assistance.
Body Bradykinesia and Hypokinesia | 1 day: Test is done once with DBS in Off state.
  Unified Parkinson's Disease Rating Scale Section III (motor examination). Combination of slowness, hesitancy, decreased arm swing, small amplitude, and poverty of movement in general. Score ranges from 0-4 where 0 is normal and 4 is unable to stand without assistance.

CONTACTS AND LOCATIONS:
Overall Officials: Hector R Martinez, MD, PhD, Principal Investigator — Hospital Zambrano Hellion
Locations (1):
- Instituto de Neurologia y Neurocirugia Hospital Zambrano Hellion, San Pedro Garza García, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ceseracciu E, Sawacha Z, Cobelli C. Comparison of markerless and marker-based motion capture technologies through simultaneous data collection during gait: proof of concept. PLoS One. 2014 Mar 4;9(3):e87640. doi: 10.1371/journal.pone.0087640. eCollection 2014. PMID 24595273
- [Background] Rocha AP, Choupina H, Fernandes JM, Rosas MJ, Vaz R, Silva Cunha JP. Parkinson's disease assessment based on gait analysis using an innovative RGB-D camera system. Annu Int Conf IEEE Eng Med Biol Soc. 2014;2014:3126-9. doi: 10.1109/EMBC.2014.6944285. PMID 25570653
- [Background] Fry AC, Herda TJ, Sterczala AJ, Cooper MA, Andre MJ. Validation of a motion capture system for deriving accurate ground reaction forces without a force plate. Big Data Anal. 2016;1(1):11. doi:10.1186/s41044-016-0008-y.
- [Background] Moodie P. Validation : Reviewing 3D Motion Capture Technology Types and What the Gold Standard Should Be for Human Movement . Lenexa, Kansas
- [Background] Rosengarden S, Docking S, Wassom D, Moodie N. The long term repeatability of a 3D markerless motion capture system and the implications it has on healthcare. J Appl Hum Mov. 2015;1(1):21-25.
- [Background] Wassom D, Fry A, Moodie N. Repeatability of 3D markerless motion capture and how it could affect between-session variability. J Appl Hum Mov. 2015;1(1):21-25.
- [Background] Mündermann L, Anguelov D, Corazza S, Chaudhari AM, Andriacchi TP. Validation of a markerless motion capture system for the calculation of lower extremity kinematics.; 2005.
- [Background] Chen SW, Lin SH, Liao LD, Lai HY, Pei YC, Kuo TS, Lin CT, Chang JY, Chen YY, Lo YC, Chen SY, Wu R, Tsang S. Quantification and recognition of parkinsonian gait from monocular video imaging using kernel-based principal component analysis. Biomed Eng Online. 2011 Nov 10;10:99. doi: 10.1186/1475-925X-10-99. PMID 22074315
- [Background] Perrott MA, Pizzari T, Cook J, McClelland JA. Comparison of lower limb and trunk kinematics between markerless and marker-based motion capture systems. Gait Posture. 2017 Feb;52:57-61. doi: 10.1016/j.gaitpost.2016.10.020. Epub 2016 Oct 31. PMID 27871019
- [Background] Galna B, Barry G, Jackson D, Mhiripiri D, Olivier P, Rochester L. Accuracy of the Microsoft Kinect sensor for measuring movement in people with Parkinson's disease. Gait Posture. 2014 Apr;39(4):1062-8. doi: 10.1016/j.gaitpost.2014.01.008. Epub 2014 Jan 22. PMID 24560691
- [Background] Bovonsunthonchai S, Vachalathiti R, Pisarnpong A, Khobhun F, Hiengkaew V. Spatiotemporal gait parameters for patients with Parkinson's disease compared with normal individuals. Physiother Res Int. 2014 Sep;19(3):158-65. doi: 10.1002/pri.1579. Epub 2013 Dec 23. PMID 24375990
- [Background] Ferrarin M, Rizzone M, Bergamasco B, Lanotte M, Recalcati M, Pedotti A, Lopiano L. Effects of bilateral subthalamic stimulation on gait kinematics and kinetics in Parkinson's disease. Exp Brain Res. 2005 Jan;160(4):517-27. doi: 10.1007/s00221-004-2036-5. Epub 2004 Oct 22. PMID 15502989
- [Background] Dewey DC, Miocinovic S, Bernstein I, Khemani P, Dewey RB 3rd, Querry R, Chitnis S, Dewey RB Jr. Automated gait and balance parameters diagnose and correlate with severity in Parkinson disease. J Neurol Sci. 2014 Oct 15;345(1-2):131-8. doi: 10.1016/j.jns.2014.07.026. Epub 2014 Jul 19. PMID 25082782
- [Background] Espy DD, Yang F, Bhatt T, Pai YC. Independent influence of gait speed and step length on stability and fall risk. Gait Posture. 2010 Jul;32(3):378-82. doi: 10.1016/j.gaitpost.2010.06.013. Epub 2010 Jul 23. PMID 20655750